CLINICAL TRIAL: NCT00142675
Title: Using Peers to Promote Exercise in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 254; R01HL072489 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical Activity

SUMMARY:
A randomized controlled trial to evaluate the effects of a 12-month telephone-supervised, home-based physical activity intervention, delivered via health educators versus supervised, trained peers, on physical activity patterns. Inactive men and women ages 50 years and older will be randomly assigned to one of these two programs or to an attention-control arm.

DETAILED DESCRIPTION:
BACKGROUND:

Despite the recognized benefits of regular physical activity, older adults remain among the most inactive segments of the U.S. population. A number of studies have demonstrated the health impact and resultant reduction in chronic disease risk achieved by improving physical activity patterns. Effective telephone-based counseling approaches for promoting and sustaining regular physical activity among older adults have been developed and validated. Such mediated interventions provide a level of individual tailoring and ongoing support to long-term adherence, while allowing for ongoing program delivery that is more flexible, convenient, and potentially lower-cost than face-to face program delivery formats. Telephone-based delivery format also allows for potentially greater reach into segments of the older population that may find it difficult or unappealing to come to community settings on a regular basis.

DESIGN NARRATIVE:

A 12-month randomized trial in which women and men ages 50 years and above living in the San Francisco Bay area who meet medical and physical activity criteria, following a baseline evaluation, be randomized to one of three study arms: telephone-supervised, home-based physical activity instruction via a trained health educator; telephone-supervised, home-based physical activity instruction via a supervised peer facilitator; or an attention-control arm consisting of health educator-based telephone delivery of non-physical activity oriented health information and support. All subjects will have a follow-up evaluation at 6 and 12 months.

ELIGIBILITY:
Women and men ages 50 years and above of the San Francisco Bay area who are free of any medical condition or disorder that would limit participation in moderate intensity exercise, not hypertensive, stable on all medications, possess English-speaking and reading skills, and are available and able to participate in the evaluations and intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)